CLINICAL TRIAL: NCT06154395
Title: A Comparative Study of 60 MHz HD-IVUS, OCT, and Conventional Angiography to Guide Reperfusion Therapy for Improving Myocardial Microcirculation Dysfunction After Acute Anterior Myocardial Infarction
Brief Title: Study on the Improvement of Myocardial Microcirculation After Acute Anterior Myocardial Infarction
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Harbin Medical University (Other)
Responsible Party: Principal Investigator, Yu Bo, Director of Department of Cardiology, Harbin Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: KY2023-137
Record Dates: First submitted 2023-11-23; First posted 2023-12-04 (Actual); Last update posted 2024-10-18 (Actual); Status verified 2024-10

CONDITIONS: Intravascular Imaging and Microvascular Obstruction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- OCT-guided group (Experimental)
  Interventions: Procedure: OCT-guided PCI
- 60 MHz HD-IVUS-guided group (Experimental)
  Interventions: Procedure: 60 MHz HD-IVUS-guided PCI
- Angiography-guided group (Active Comparator)
  Interventions: Procedure: Angiography-guided PCI

INTERVENTIONS:
Procedure: OCT-guided PCI — The OCT guidance team routinely conducts OCT examinations on patients after standard angiography and/or thrombus aspiration. The OCT examination follows a standard procedure. The operator evaluates the stability of the lesion and decides whether to proceed with stent implantation therapy (with the option to choose the type of stent) or opt for conservative medical treatment. If a stent is implanted, the procedure is carried out according to guidelines and standard protocols, with the landing zone of the stent determined based on OCT image features. After stent implantation, a follow-up OCT examination of the stent segment, as well as angiographic examination, is performed. Based on the OCT results, the operator decides whether post-dilation is necessary.
  Arms: OCT-guided group
Procedure: 60 MHz HD-IVUS-guided PCI — The IVUS guidance team routinely conducts IVUS examinations on patients after standard angiography and/or thrombus aspiration. The IVUS examination follows a standard procedure. The operator evaluates the stability of the lesion and decides whether to proceed with stent implantation therapy (with the option to choose the type of stent) or opt for conservative medical treatment. If a stent is implanted, the procedure is carried out according to guidelines and standard protocols, with the landing zone of the stent determined based on IVUS image features. After stent implantation, a follow-up IVUS examination of the stent segment, as well as angiographic examination, is performed. Based on the IVUS results, the operator decides whether post-dilation is necessary.
  Arms: 60 MHz HD-IVUS-guided group
Procedure: Angiography-guided PCI — After routine angiography and/or thrombus aspiration, the operator assesses the lesion based on treatment standards to determine whether stent implantation is necessary. For patients undergoing stent implantation, a follow-up angiography is performed postoperatively, and the decision for post-dilation is made by the operator based on experience.
  Arms: Angiography-guided group

SUMMARY:
This study is a prospective, single-center, randomized controlled clinical trial. Ninety patients with anterior wall ST-segment elevation myocardial infarction (STEMI) who are planned for primary percutaneous coronary intervention (PCI) within 6 hours of symptom onset will be screened. Patients with inclusion criteria and without exclusion criteria will be randomized into three groups in a 1:1:1 ratio: OCT-guided group, 60 MHz HD-IVUS-guided group, and angiography-guided group after signing the informed consent form.

Based on the lesion characteristics detected by imaging in each group, coronary revascularization will be performed for the culprit vessels of myocardial infarction. The TIMI myocardial perfusion frame count (TMPFC) values of the culprit vessels will be recorded immediately after PCI, and secondary prevention medications for myocardial infarction will be administered. Three days after the procedure, a 3.0T cardiac magnetic resonance imaging (MRI) with gadolinium diethylenetriaminepentaacetic acid (Gd-DTPA) delayed enhancement (LEG) scan will be conducted to assess the microvascular obstruction (MVO) area.

Patients will be followed in the outpatient clinic visit at 1 month (with a window period of XX days) after discharge, and a repeat cardiac MRI will be performed to determine the presence of MVO and the size of the myocardial infarction.

ELIGIBILITY:
Inclusion Criteria:

Clinical Inclusion Criteria:

1. Subjects aged ≥18 years;
2. Initial diagnosis of anterior wall ST-segment elevation myocardial infarction, with symptoms occurring within 6 hours, and undergoing primarypercutaneous coronary intervention (PCI);
3. Subjects (or legal representatives) who understand the study requirements and treatment procedures and provide signed informed consent.

Imaging Inclusion Criteria (Visual Estimation):

1. Target lesion is the culprit lesion, located in the native coronary artery, with a visually estimated reference vessel diameter (RVD) between 2.25 mm and 4.0 mm;
2. Culprit segment of the infarct-related artery (IRA) is located between the origin of the left anterior descending (LAD) artery and the emergence of the second diagonal branch (D2);
3. After pre-treatment , the degree of stenosis in the LAD is ≤90%, and TIMI flow is grade 3.

Exclusion Criteria:

Clinical Exclusion Criteria:

1. History of coronary artery bypass grafting (CABG);
2. Known history of myocardial infarction or PCI;
3. Previous thrombolytic therapy before PCI;
4. Severe liver or kidney dysfunction, severe valvular heart disease, chronic obstructive pulmonary disease, etc.;
5. Contraindications to magnetic resonance imaging;
6. Allergy to gadolinium contrast agents and/or accompanying medications for devices or procedures (e.g., any component of drug-eluting stents, all P2Y12 inhibitors, or aspirin);
7. Expected lifespan of the subject less than 12 months;
8. Pregnant or lactating females;
9. Other subjects deemed unsuitable for participation in the study by the investigator.

Imaging Exclusion Criteria (Visual Estimation):

1. Presence of lesions requiring intervention other than the target lesion at baseline surgery;
2. No protected left main coronary artery disease (visual estimate of stenosis >50%);
3. Diffuse severe calcification (>20 mm) or chronic total occlusion in the major coronary vessels (LCX, RCA);
4. Severe coronary artery tortuosity (>45°) or calcification (>270°), or other conditions that may interfere with the use of intravascular imaging.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2023-12-20 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Microvascular obstruction (MVO) assessed by cardiac magnetic resonance imaging (CMR) | Three days after percutaneous coronary intervention (PCI)
  The area of microvascular obstruction (MVO) assessed by cardiac magnetic resonance imaging (CMR) three days after percutaneous coronary intervention (PCI).

CONTACTS AND LOCATIONS:
Overall Officials: Bo Yu, M.D.; Ph.D., Principal Investigator — The Second Affiliated Hospital of Harbin Medical University
Locations (1):
- The 2nd Affiliated Hospital of Harbin Medical University, Harbin, Heilongjiang, China

IPD SHARING:
Plan to Share IPD: Undecided